CLINICAL TRIAL: NCT03720652
Title: Mindful Self-Compassion Training to Improve Retention, Job Satisfaction, and Attitudes Toward Dementia Among Long-Term Care Nursing Assistants
Brief Title: Certified Nursing Assistants' Wellbeing
Acronym: CNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-2012; 1R21AG058133-01A1 (NIH)
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Results first posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-03

CONDITIONS: Stress and Burnout
Keywords: Mindfulness; Certified Nursing Assistants; Long-Term Care; Staff Turnover; Mindful Self-Compassion
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: In Aim 1, the 8-week MSC program was conducted with nursing assistants from 1 nursing home to test for feasibility and practicality.
  After receiving feedback from participants of Aim 1, in Aim 2, the MSC program will be conducted in 2 nursing homes. Both nursing homes in Aim 2 will receive a shortened 6-week, 1 hour version specific to health care staff, in order to test the feasibility and practicality.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8-Week Mindful Self-Compassion (MSC) (Experimental): CNAs in Aim 1 will participate in the standardized, 8-week Mindful Self-Compassion course. Each 8-week session will last for 2.5 hours. Also included is a half day retreat, that CNAs may attend if they are able.
  Interventions: Behavioral: 8-Week Mindful Self-Compassion (MSC)
- 6-Week Mindful Self Compassion (MSC) (Experimental): CNAs from both nursing homes in Aim 2 will participate in the 6-week Mindful Self-Compassion course, that was shortened and customized to fit the needs of health care staff. Each 6-week session will last for 1 hour.
  Interventions: Behavioral: 6-Week Mindful Self-Compassion (MSC)

INTERVENTIONS:
Behavioral: 8-Week Mindful Self-Compassion (MSC) — The 8-week MSC is a course of eight 2.5 hour weekly sessions that is based off self-compassion, a construct closely related to mindfulness. Self-compassion (SC) has three main interrelated components: self-kindness, common humanity, and mindfulness. MSC is an 8-session program that integrates SC and mindfulness.
  It includes the following components:
  * Discovering Mindful Self-Compassion
  * Practicing Mindfulness
  * Practicing Lovingkindness
  * Discovering your Compassionate Voice
  * Living Deeply
  * Meeting Difficult Emotions
  * Exploring Challenging Relationships
  * Embracing Your Life
  Arms: 8-Week Mindful Self-Compassion (MSC)
Behavioral: 6-Week Mindful Self-Compassion (MSC) — The 6-week MSC is a course of six 1 hour weekly sessions that is based off self-compassion, a construct closely related to mindfulness. Self-compassion (SC) has three main interrelated components: self-kindness, common humanity, and mindfulness. MSC is an 6-session program that integrates SC and mindfulness.
  It includes the following components:
  * What is Self-Compassion
  * Practicing Self-Compassion
  * Discovering your Compassionate Voice
  * Self-Compassion and Resilience
  * Self-Compassion and Burnout
  * Going Forward This program is a shortened version of the 8-week program, specifically created for the needs of health care staff.
  Arms: 6-Week Mindful Self Compassion (MSC)

SUMMARY:
Certified nursing assistants (CNAs), who provide the majority of care to persons with chronic disease and/or cognitive impairment from Alzheimer's disease and related dementias, face tremendous job and home stress, and as a result absenteeism and job turnover are high. This is a preliminary study that will tailor Mindful Self-Compassion (MSC) - a promising new program designed to cultivate greater self-care, and strengthen resilience and coping skills - for the CNA population and study its effectiveness. If results are favorable, MSC could be incorporated into CNA training programs, thereby helping contribute to a more effective and stable long-term care workforce.

DETAILED DESCRIPTION:
U.S. nursing homes (NHs) serve 1.6 million older persons, all of whom have significant physical and/or cognitive impairment, and the majority of whom have Alzheimer's disease or a related cognitive disorder. In these settings the vast majority of hands-on care is provided by an estimated 634,000 certified nursing assistants (CNAs) - paraprofessional caregivers who are racially diverse, largely female, and an annual income equivalent to the poverty threshold for a family of four. Despite the crucial role of CNAs in providing care for the long-term care population and efforts to recruit and retain a stable workforce, absenteeism rates are high and annual turnover averages 65%, with adverse impact on the quality of care provided to NH residents, making CNA retention a policy priority.

CNAs have significant life stressors that affect their ability to work, such as single parenthood, poor physical health, difficulty finding childcare, and transportation problems. They also face emotionally and physically demanding job tasks, particularly when working with persons with Alzheimer's disease and related dementias, and many lack helpful strategies for dealing with stress, negative feelings, and burden.

A newly developed, standardized Mindful Self-Compassion (MSC) intervention may have particularly high impact and relevance for the high-stress lives of NH CNAs. MSC training has been shown to increase wellbeing, compassion for others, and stress-coping skills. However, little is known about the impact, feasibility and acceptability of MSC training in low-educated, stress-burdened paraprofessional populations such as CNAs, or whether it can impact outcomes such as burnout, absenteeism, and turnover.

This preliminary study will modify, refine, and test a MSC training intervention for CNAs, to be known as the CNA Wellbeing Program, who care for nursing home residents. The researcher teams' goal is to increase CNA coping skills and well-being, thereby reducing intent to leave the job, reducing burnout, and improving job satisfaction and attitudes toward people with dementia. The proposed research will be conducted in 3 similarly rated and structured community NHs. In Aim 1 the investigators will assess intervention feasibility and acceptability in one NH, using the knowledge they gain to tailor an evidence-based MSC program specifically for CNAs. In Aim 2 the investigators will pilot test the MSC training program with 30 CNAs who work in 2 similarly rated and structured NHs, evaluating the fidelity of the revised training and exploring trends in immediate, 3-month, and 6-month outcome measures in order to inform power calculations for future trials.

The specific aims are:

Aim 1. Determine the feasibility, acceptability, and necessary adaptations of MSC training needed to meet the diverse cultural background, limited literacy, and job and family challenges of the nursing home CNA workforce, including the unique challenges of caring for persons with dementia, and of the data collection methods.

1. Conduct a field trial of the standardized 8-week MSC training program with 15 CNAs within a single community NH. Evaluation will focus on: (a) participation (including home practice adherence); (b) attendee evaluation of the training; (c) barriers to and facilitators of participation; (d) use and retention of class material by participants; and (e) recommendations for improvement of training.
2. Field test the feasibility and acceptability of our study recruitment and evaluation strategy.
3. Use data collected from the field test to modify recruitment strategies, protocols, and course structure, content and materials so as to be maximally feasible, acceptable and effective in a CNA population.

Aim 2. Conduct a pilot test of the adapted protocols and intervention in a sample of 30 CNAs from 2 similarly rated and structured community NHs to reexamine feasibility and acceptability, identify trends in key intermediate and long-term outcomes, and estimate effect size in preparation for a future randomized trial.

1. Evaluate the fidelity and immediate impact of the modified training by measuring (a) training attendance; (b) satisfaction with the training; and (c) pre-and post-training measures of self-compassion, perceived stress, job satisfaction, job burnout symptoms, and attitudes towards persons with dementia.
2. Evaluate the sustained impact of the training by comparing baseline, 3-and 6-month post-training measurements of: intent to leave job, self-compassion, perceived stress, job satisfaction, job burnout symptoms, and attitudes towards persons with dementia.

ELIGIBILITY:
Inclusion Criteria:

* Certified Nursing Assistant employed by one of 3 study Nursing Homes
* Aged 18 and over
* Speak English
* Work at least 20 hours as a CNA at one of our proposed Nursing Homes
* Expect to attend at least 75% of the intervention classes
* Expect to stay at least the course of the intervention on the job
* Score in the top 50% on the PSS-10 (Perceived Stress Scale) (if more than 20 participants interested)

Exclusion Criteria:

* Younger than 18
* Working fewer than 20 hours a week
* Unable to attend at least 75% of the intervention classes
* Expect to leave their position during the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip D Sloane, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be shared beginning 9 to 36 months following publication, and will be available for up to 7 years post publication.
Access Criteria: To access, interested parties will have to email Drs. Christine Lathren, lathren@email.unc.edu, and Philip D. Sloane, philip_sloane@med.unc.edu, or contact the study team through the Cecil G. Sheps Center for Health Services Research at (919) 966-5011.

REFERENCES:
- [Background] Jones AL, Dwyer LL, Bercovitz AR, Strahan GW. The National Nursing Home Survey: 2004 overview. Vital Health Stat 13. 2009 Jun;(167):1-155. PMID 19655659
- [Background] Barbarotta L. Direct Care Worker Retention: Strategies for Success.; 2010.
- [Background] Castle NG, Ferguson-Rome JC. Influence of Nurse Aide Absenteeism on Nursing Home Quality. Gerontologist. 2015 Aug;55(4):605-15. doi: 10.1093/geront/gnt167. Epub 2014 Jan 7. PMID 24398653
- [Background] Castle NG, Engberg J, Men A. Nursing home staff turnover: impact on nursing home compare quality measures. Gerontologist. 2007 Oct;47(5):650-61. doi: 10.1093/geront/47.5.650. PMID 17989407
- [Background] Lerner NB, Johantgen M, Trinkoff AM, Storr CL, Han K. Are nursing home survey deficiencies higher in facilities with greater staff turnover. J Am Med Dir Assoc. 2014 Feb;15(2):102-7. doi: 10.1016/j.jamda.2013.09.003. Epub 2013 Oct 15. PMID 24139163
- [Background] Trinkoff AM, Han K, Storr CL, Lerner N, Johantgen M, Gartrell K. Turnover, staffing, skill mix, and resident outcomes in a national sample of US nursing homes. J Nurs Adm. 2013 Dec;43(12):630-6. doi: 10.1097/NNA.0000000000000004. PMID 24232236
- [Background] Cook G, Brown-Wilson C. Care home residents' experiences of social relationships with staff. Nurs Older People. 2010 Feb;22(1):24-9. doi: 10.7748/nop2010.02.22.1.24.c7492. PMID 20225727
- [Background] Squillace MR, Remsburg RE, Harris-Kojetin LD, Bercovitz A, Rosenoff E, Han B. The National Nursing Assistant Survey: improving the evidence base for policy initiatives to strengthen the certified nursing assistant workforce. Gerontologist. 2009 Apr;49(2):185-97. doi: 10.1093/geront/gnp024. Epub 2009 Apr 1. PMID 19363014
- [Background] Dill JS, Morgan JC, Marshall VW, Pruchno R. Contingency, employment intentions, and retention of vulnerable low-wage workers: an examination of nursing assistants in nursing homes. Gerontologist. 2013 Apr;53(2):222-34. doi: 10.1093/geront/gns085. Epub 2012 Aug 8. PMID 22875015
- [Background] Lachs MS, Rosen T, Teresi JA, Eimicke JP, Ramirez M, Silver S, Pillemer K. Verbal and physical aggression directed at nursing home staff by residents. J Gen Intern Med. 2013 May;28(5):660-7. doi: 10.1007/s11606-012-2284-1. Epub 2012 Dec 8. PMID 23225256
- [Background] Chappell NL, Novak M. Caring for institutionalized elders: Stress among nursing assistants. J Appl Gerontol. 1994;13(3):299-315.
- [Background] Morgan DG, Stewart NJ, D'Arcy C, Forbes D, Lawson J. Work stress and physical assault of nursing aides in rural nursing homes with and without dementia special care units. J Psychiatr Ment Health Nurs. 2005 Jun;12(3):347-58. doi: 10.1111/j.1365-2850.2005.00846.x. PMID 15876243
- [Background] Schaefer JA, Moos RH. Effects of work stressors and work climate on long-term care staff's job morale and functioning. Res Nurs Health. 1996 Feb;19(1):63-73. doi: 10.1002/(SICI)1098-240X(199602)19:13.0.CO;2-J. PMID 8552804
- [Background] Cooper SL, Carleton HL, Chamberlain SA, Cummings GG, Bambrick W, Estabrooks CA. Burnout in the nursing home health care aide: A systematic review. Burn Res. 2016;3:76-87.
- [Background] Astrom S, Nilsson M, Norberg A, Sandman PO, Winblad B. Staff burnout in dementia care--relations to empathy and attitudes. Int J Nurs Stud. 1991;28(1):65-75. doi: 10.1016/0020-7489(91)90051-4. PMID 1856035
- [Background] Moyle W, Murfield JE, Griffiths SG, Venturato L. Care staff attitudes and experiences of working with older people with dementia. Australas J Ageing. 2011 Dec;30(4):186-90. doi: 10.1111/j.1741-6612.2010.00470.x. Epub 2010 Oct 8. PMID 22176562
- [Background] Zimmerman S, Williams CS, Reed PS, Boustani M, Preisser JS, Heck E, Sloane PD. Attitudes, stress, and satisfaction of staff who care for residents with dementia. Gerontologist. 2005 Oct;45 Spec No 1(1):96-105. doi: 10.1093/geront/45.suppl_1.96. PMID 16230756
- [Background] Bauer-Wu S, Fontaine D. Prioritizing Clinician Wellbeing: The University of Virginia's Compassionate Care Initiative. Glob Adv Health Med. 2015 Sep;4(5):16-22. doi: 10.7453/gahmj.2015.042. Epub 2015 Sep 1. PMID 26421230
- [Background] Bodenheimer T, Sinsky C. From triple to quadruple aim: care of the patient requires care of the provider. Ann Fam Med. 2014 Nov-Dec;12(6):573-6. doi: 10.1370/afm.1713. PMID 25384822
- [Background] Kabat-Zinn J. Wherever You Go, There You Are: Mindfulness in Everyday Life. New York: Hyperion; 1994.
- [Background] Khoury B, Sharma M, Rush SE, Fournier C. Mindfulness-based stress reduction for healthy individuals: A meta-analysis. J Psychosom Res. 2015 Jun;78(6):519-28. doi: 10.1016/j.jpsychores.2015.03.009. Epub 2015 Mar 20. PMID 25818837
- [Background] Gotink RA, Chu P, Busschbach JJ, Benson H, Fricchione GL, Hunink MG. Standardised mindfulness-based interventions in healthcare: an overview of systematic reviews and meta-analyses of RCTs. PLoS One. 2015 Apr 16;10(4):e0124344. doi: 10.1371/journal.pone.0124344. eCollection 2015. PMID 25881019 (Retraction: PMID 30978236 PLoS One. 2019 Apr 12;14(4):e0215608)
- [Background] Li G, Yuan H, Zhang W. The Effects of Mindfulness-Based Stress Reduction for Family Caregivers: Systematic Review. Arch Psychiatr Nurs. 2016 Apr;30(2):292-9. doi: 10.1016/j.apnu.2015.08.014. Epub 2015 Aug 28. PMID 26992885
- [Background] Irving JA, Dobkin PL, Park J. Cultivating mindfulness in health care professionals: a review of empirical studies of mindfulness-based stress reduction (MBSR). Complement Ther Clin Pract. 2009 May;15(2):61-6. doi: 10.1016/j.ctcp.2009.01.002. Epub 2009 Feb 28. PMID 19341981
- [Background] Lamothe M, Rondeau E, Malboeuf-Hurtubise C, Duval M, Sultan S. Outcomes of MBSR or MBSR-based interventions in health care providers: A systematic review with a focus on empathy and emotional competencies. Complement Ther Med. 2016 Feb;24:19-28. doi: 10.1016/j.ctim.2015.11.001. Epub 2015 Nov 27. PMID 26860797
- [Background] Smith SA. Mindfulness-based stress reduction: an intervention to enhance the effectiveness of nurses' coping with work-related stress. Int J Nurs Knowl. 2014 Jun;25(2):119-30. doi: 10.1111/2047-3095.12025. Epub 2014 Feb 26. PMID 24612607
- [Background] Cohen-Katz J, Wiley SD, Capuano T, Baker DM, Kimmel S, Shapiro S. The effects of mindfulness-based stress reduction on nurse stress and burnout, Part II: A quantitative and qualitative study. Holist Nurs Pract. 2005 Jan-Feb;19(1):26-35. doi: 10.1097/00004650-200501000-00008. PMID 15736727
- [Background] Mackenzie CS, Poulin PA, Seidman-Carlson R. A brief mindfulness-based stress reduction intervention for nurses and nurse aides. Appl Nurs Res. 2006 May;19(2):105-9. doi: 10.1016/j.apnr.2005.08.002. PMID 16728295
- [Background] Baker C, Huxley P, Dennis M, Islam S, Russell I. Alleviating staff stress in care homes for people with dementia: protocol for stepped-wedge cluster randomised trial to evaluate a web-based Mindfulness- Stress Reduction course. BMC Psychiatry. 2015 Dec 21;15:317. doi: 10.1186/s12888-015-0703-7. PMID 26691663
- [Background] Zeller JM, Lamb K. Mindfulness meditation to improve care quality and quality of life in long-term care settings. Geriatr Nurs. 2011 Mar-Apr;32(2):114-8. doi: 10.1016/j.gerinurse.2010.11.006. Epub 2011 Jan 15. PMID 21239085
- [Background] Raab K. Mindfulness, self-compassion, and empathy among health care professionals: a review of the literature. J Health Care Chaplain. 2014;20(3):95-108. doi: 10.1080/08854726.2014.913876. PMID 24926896
- [Background] Egan H, Mantzios M, Jackson C. Health Practitioners and the Directive Towards Compassionate Healthcare in the UK: Exploring the Need to Educate Health Practitioners on How to be Self-Compassionate and Mindful Alongside Mandating Compassion Towards Patients. Heal Prof Educ. 2016:9-11.
- [Background] Neff KD, Dahm KA. Self-Compassion: What It Is, What It Does, and How It Relates to Mindfulness. (Robinson M, Meier B, Ostafin B, eds.). New York: Springer; 2015.
- [Background] Zessin U, Dickhauser O, Garbade S. The Relationship Between Self-Compassion and Well-Being: A Meta-Analysis. Appl Psychol Health Well Being. 2015 Nov;7(3):340-64. doi: 10.1111/aphw.12051. Epub 2015 Aug 26. PMID 26311196
- [Background] MacBeth A, Gumley A. Exploring compassion: a meta-analysis of the association between self-compassion and psychopathology. Clin Psychol Rev. 2012 Aug;32(6):545-52. doi: 10.1016/j.cpr.2012.06.003. Epub 2012 Jun 23. PMID 22796446
- [Background] Leary MR, Tate EB, Adams CE, Allen AB, Hancock J. Self-compassion and reactions to unpleasant self-relevant events: the implications of treating oneself kindly. J Pers Soc Psychol. 2007 May;92(5):887-904. doi: 10.1037/0022-3514.92.5.887. PMID 17484611
- [Background] Wiklund Gustin L, Wagner L. The butterfly effect of caring - clinical nursing teachers' understanding of self-compassion as a source to compassionate care. Scand J Caring Sci. 2013 Mar;27(1):175-83. doi: 10.1111/j.1471-6712.2012.01033.x. Epub 2012 Jun 27. PMID 22734628
- [Background] Mills J, Wand T, Fraser JA. On self-compassion and self-care in nursing: selfish or essential for compassionate care? Int J Nurs Stud. 2015 Apr;52(4):791-3. doi: 10.1016/j.ijnurstu.2014.10.009. Epub 2014 Oct 25. No abstract available. PMID 25457876
- [Background] Gerber Z, Tolmacz R, Doron Y. Self-compassion and forms of concern for others. Pers Individ Dif. 2015;86:394-400.
- [Background] Duarte J, Pinto-Gouveia J, Cruz B. Relationships between nurses' empathy, self-compassion and dimensions of professional quality of life: A cross-sectional study. Int J Nurs Stud. 2016 Aug;60:1-11. doi: 10.1016/j.ijnurstu.2016.02.015. Epub 2016 Mar 4. PMID 27297364
- [Background] Durkin M, Beaumont E, Hollins Martin CJ, Carson J. A pilot study exploring the relationship between self-compassion, self-judgement, self-kindness, compassion, professional quality of life and wellbeing among UK community nurses. Nurse Educ Today. 2016 Nov;46:109-114. doi: 10.1016/j.nedt.2016.08.030. Epub 2016 Aug 30. PMID 27621200
- [Background] Beaumont E, Durkin M, Hollins Martin CJ, Carson J. Compassion for others, self-compassion, quality of life and mental well-being measures and their association with compassion fatigue and burnout in student midwives: A quantitative survey. Midwifery. 2016 Mar;34:239-244. doi: 10.1016/j.midw.2015.11.002. Epub 2015 Nov 6. PMID 26628352
- [Background] Neff KD, Germer CK. A pilot study and randomized controlled trial of the mindful self-compassion program. J Clin Psychol. 2013 Jan;69(1):28-44. doi: 10.1002/jclp.21923. Epub 2012 Oct 15. PMID 23070875
- [Background] Bluth K, Gaylord SA, Campo RA, Mullarkey MC, Hobbs L. Making Friends With Yourself: A Mixed Methods Pilot Study of a Mindful Self-Compassion Program for Adolescents. Mindfulness (N Y). 2016 Mar 1;7(2):479-492. doi: 10.1007/s12671-015-0476-6. Epub 2015 Dec 19. PMID 27110301
- [Background] Bluth K, Eisenlohr-Moul TA. Response to a mindful self-compassion intervention in teens: A within-person association of mindfulness, self-compassion, and emotional well-being outcomes. J Adolesc. 2017 Jun;57:108-118. doi: 10.1016/j.adolescence.2017.04.001. Epub 2017 Apr 14. PMID 28414965
- [Background] Friis AM, Johnson MH, Cutfield RG, Consedine NS. Kindness Matters: A Randomized Controlled Trial of a Mindful Self-Compassion Intervention Improves Depression, Distress, and HbA1c Among Patients With Diabetes. Diabetes Care. 2016 Nov;39(11):1963-1971. doi: 10.2337/dc16-0416. Epub 2016 Jun 22. PMID 27335319
- [Background] McPherson S, Hiskey S, Alderson Z. Distress in working on dementia wards - A threat to compassionate care: A grounded theory study. Int J Nurs Stud. 2016 Jan;53:95-104. doi: 10.1016/j.ijnurstu.2015.08.013. Epub 2015 Sep 3. PMID 26384957
- [Background] Allen AB, Leary MR. Self-Compassion, Stress, and Coping. Soc Personal Psychol Compass. 2010 Feb 1;4(2):107-118. doi: 10.1111/j.1751-9004.2009.00246.x. PMID 20686629
- [Background] Abercrombie PD, Zamora A, Korn AP. Lessons learned: providing a mindfulness-based stress reduction program for low-income multiethnic women with abnormal pap smears. Holist Nurs Pract. 2007 Jan-Feb;21(1):26-34. doi: 10.1097/00004650-200701000-00006. PMID 17167329
- [Background] Lee EH. Review of the psychometric evidence of the perceived stress scale. Asian Nurs Res (Korean Soc Nurs Sci). 2012 Dec;6(4):121-7. doi: 10.1016/j.anr.2012.08.004. Epub 2012 Sep 18. PMID 25031113
- [Background] Rosen J, Stiehl EM, Mittal V, Leana CR. Stayers, leavers, and switchers among certified nursing assistants in nursing homes: a longitudinal investigation of turnover intent, staff retention, and turnover. Gerontologist. 2011 Oct;51(5):597-609. doi: 10.1093/geront/gnr025. Epub 2011 Apr 15. PMID 21498629
- [Background] Sloane PD, Williams CS, Zimmerman S. Immigrant status and intention to leave of nursing assistants in U.S. nursing homes. J Am Geriatr Soc. 2010 Apr;58(4):731-7. doi: 10.1111/j.1532-5415.2010.02781.x. PMID 20398155
- [Background] Cohen S, Williamson G. The social psychology of health: Claremont symposium on applied social psychology. In: Perceived Stress in a Probability Sample of the United States. In: Spacapan S, Oskamp S, Eds. Newbury Park, CA: Sage; 1988.
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Roberti J, Harrington L, Storch E. Further psychometric support for the 10- item version of the perceived stress scale. J Coll Couns. 2006;9(2):135-147.
- [Background] Lintern T, Woods B, Phair L. Training is not enough to change care practice. J Dement Care. 2000;8:15-17.
- [Background] Lintern T. Quality in Dementia Care: Evaluating Staff Attitudes and Behaviour. 2001.
- [Background] Kada S, Nygaard HA, Mukesh BN, Geitung JT. Staff attitudes towards institutionalised dementia residents. J Clin Nurs. 2009 Aug;18(16):2383-92. doi: 10.1111/j.1365-2702.2009.02791.x. PMID 19583668
- [Background] Maslach C, Jackson S, Leiter M. Maslach Burnout Inventory. Palo Alto; 1986.
- [Background] Rafferty JP, Lemkau JP, Purdy RR, Rudisill JR. Validity of the Maslach Burnout Inventory for family practice physicians. J Clin Psychol. 1986 May;42(3):488-92. doi: 10.1002/1097-4679(198605)42:33.0.co;2-s. PMID 3711351
- [Background] Schaufeli WB, Bakker AB, Hoogduin K, Schaap C, Kladler A. on the clinical validity of the maslach burnout inventory and the burnout measure. Psychol Health. 2001 Sep;16(5):565-82. doi: 10.1080/08870440108405527. PMID 22804499
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Diener E, Inglehart R, Tay L. Theory and validity of life satisfaction scales. Soc Indic Res. 2013;112(3):497-527.
- [Background] Cammann C, Fichman M, Jenkins D, Klesh J. Assessing the attitudes and perceptions of organizational members. In: Assessing Organizational Change: A Guide to Methods, Measures, and Practices. Vol 71.; 1983.
- [Background] McFarlin D, Rice R. The role of facet importance as a moderator in job satisfaction processes. J Organ Behav. 1992;13(1):41-54.
- [Background] Pearson C. An assessment of extrinsic feedback on participation, role perceptions, motivation, and job satisfaction in a self-managed system for monitoring group achievement. Hum relations.1991;44(5):517-537.
- [Background] Sanchez J, Brock P. Sanchez JI, Brock P. Outcomes of perceived discrimination among Hispanic employees: is diversity management a luxury or a necessity? Academy of Management Journal. 1996;39(3):704-719. Acad Manag Journal. 1996;39(3):704-719.
- [Background] Siegall M, McDonald T. Focus of Attention and Employee Reactions to Job Change. J Appl Soc Psychol. 1995;25(13):1121-1141.
- [Background] McLain DL. Responses to health and safety risk in the work environment. Acad Manage J. 1995 Dec;38(6):1726-43. PMID 10169684
- [Background] Sanchez J, Kraus E, White S, Williams M. Adopting high-involvement human resource practices the mediating role of benchmarking. Gr Organ Manag. 1999;24(4):461-478.
- [Background] George J. Leader positive mood and group performance: The case of customer service. J Appl Soc Psychol. 1995;25(9):778-794.
- [Background] Fletcher S, Zimmerman S, Preisser JS, Mitchell C, Reed D, Gould E, Beeber A, Reed P. Implementation fidelity of a standardized Dementia Care training program across multiple trainers and settings. Alzheimers care today. 2010;11(1):51-60.
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- See also: Nursing Home Compare — https://www.medicare.gov/nursinghomecompare/search.html
- See also: Unscheduled Absence Survey: CCH Survey Finds Unscheduled Absenteeism Up in U.S. Workplaces. — http://www.cch.com/press/news/2006/20061026h.asp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from all three nursing homes were recruited between March of 2019 and October of 2019. Participants from Nursing Home 1 were recruited in March/April 2019 and participants from Nursing Homes 2 & 3 were recruited in September/October of 2019. Recruitment took place on-site at each nursing home, during staff meetings and shift changes.
Groups:
- 8-Week Mindful Self-Compassion (MSC): CNAs in Aim 1 will participate in the standardized, 8-week Mindful Self-Compassion course. Each 8-week session will last for 2.5 hours.
  8-Week Mindful Self-Compassion (MSC): The 8-week MSC is a course of eight 2.5 hour weekly sessions that is based off self-compassion, a construct closely related to mindfulness. Self-compassion (SC) has three main interrelated components: self-kindness, common humanity, and mindfulness. MSC is an 8-session program that integrates SC and mindfulness.
  It includes the following components:
  * Discovering Mindful Self-Compassion
  * Practicing Mindfulness
  * Practicing Lovingkindness
  * Discovering your Compassionate Voice
  * Living Deeply
  * Meeting Difficult Emotions
  * Exploring Challenging Relationships
  * Embracing Your Life
- 6-Week Mindful Self Compassion (MSC): CNAs from both nursing homes in Aim 2 will participate in the 6-week Mindful Self-Compassion course, that was shortened and customized to fit the needs of health care staff. Each 6-week session will last for 1 hour.
  6-Week Mindful Self-Compassion (MSC): The 6-week MSC is a course of six 1 hour weekly sessions that is based off self-compassion, a construct closely related to mindfulness. Self-compassion (SC) has three main interrelated components: self-kindness, common humanity, and mindfulness. MSC is an 6-session program that integrates SC and mindfulness.
  It includes the following components:
  * What is Self-Compassion
  * Practicing Self-Compassion
  * Discovering your Compassionate Voice
  * Self-Compassion and Resilience
  * Self-Compassion and Burnout
  * Going Forward
  This program is a shortened version of the 8-week program, specifically created for the needs of health care staff.
Period: Overall Study
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Started (# of Participants to Complete Screening Questionnaire) | 12 | 27
Baseline Interview (# Participants to Complete Baseline Interview) | 12 | 22
Start Intervention (# of Participants to Start Intervention (i.e. attend at least one intervention session)) | 11 | 21
Complete Intervention (# of Participants to Finish Intervention (i.e. attend throughout intervention)) | 10 | 20
3-Month Follow Up Interview (# Participants to Complete 3-Month Follow Up Interview) | 10 | 19
6-Month Follow Up Interview (# Participants to Complete 6-Month Follow Up Interview) | 10 | 16
Completed | 10 | 16
Not Completed | 2 | 11
Not completed — Withdrawal by Subject | 2 | 7
Not completed — Lost to Follow-up | 0 | 4

BASELINE CHARACTERISTICS:
Population: Analysis population is composed of participants who began intervention.
Groups:
- 8-Week Mindful Self-Compassion (MSC): CNAs in Aim 1 participated in the standardized, 8-week Mindful Self-Compassion course. Each 8-week session lasted for 2.5 hours.
- 6-Week Mindful Self Compassion (MSC): CNAs from both nursing homes in Aim 2 participated in the 6-week Mindful Self-Compassion course, that was shortened and customized to fit the needs of health care staff.
- Total: Total of all reporting groups
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC) | Total
Number analyzed (Participants) | 11 | 21 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Analysis population includes participants for whom year of birth was gathered.
  years
    number analyzed (Participants) | 10 | 20 | 30
    (all) | 47.70 (11.42) | 50.40 (10.01) | 49.50 (10.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 19 | 30
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 17 | 23
  Unknown or Not Reported | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 9 | 18 | 27
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Study Participant's Self-Rating of Likelihood to Leave Job in the Coming Year Over Time
Description: The researchers will assess intent to leave job by asking "How likely is it that you will leave this job in the next year? "Would you say... 1 is Not at All Likely, 2 is Somewhat Likely, 3 is Very Likely." Minimum = 1 (best value), maximum = 3 (worst value). For the primary outcome analysis, intent will be evaluated by totaling the count of participants who responded "Somewhat Likely", "Very likely", or "Not at all likely." This was collected over the course of four time frames: Baseline, End-of Intervention interview, 3-Month Follow Up Interview, and 6-Month Follow Up Interview.
Time Frame: Participants will be followed for the duration of the intervention and 6 additional months after the intervention ends, an expected average of 8 months
Population: Analysis population is composed of participants who began the intervention. All collected data are reported. Some data are missing due to study attrition or nonresponse.
Measure: Count of Participants; unit: Participants
Groups:
- 8-Week Mindful Self-Compassion (MSC): CNAs in Aim 1 will participate in the standardized, 8-week Mindful Self-Compassion course. Each 8-week session will last for 2.5 hours.
- 6-Week Mindful Self Compassion (MSC): CNAs from both nursing homes in Aim 2 will participate in the 6-week Mindful Self-Compassion course, that was shortened and customized to fit the needs of health care staff.
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Number analyzed (Participants) | 11 | 21
Participants
  Baseline: Not at All Likely to Leave Job | 9 | 13
  Baseline: Somewhat Likely to Leave Job | 1 | 5
  Baseline: Very Likely to Leave Job | 1 | 3
  End-of-Intervention Interview: number analyzed (Participants) | 10 | 20
  End-of-Intervention Interview: Not at All Likely to Leave Job | 6 | 9
  End-of-Intervention Interview: Somewhat Likely to Leave Job | 2 | 8
  End-of-Intervention Interview: Very Likely to Leave Job | 2 | 3
  3-Month Follow Up Interview: number analyzed (Participants) | 9 | 18
  3-Month Follow Up Interview: Not at All Likely to Leave Job | 6 | 8
  3-Month Follow Up Interview: Somewhat Likely to Leave Job | 2 | 7
  3-Month Follow Up Interview: Very Likely to Leave Job | 1 | 3
  6-Month Follow Up Interview: number analyzed (Participants) | 7 | 16
  6-Month Follow Up Interview: Not at All Likely to Leave Job | 6 | 6
  6-Month Follow Up Interview: Somewhat Likely to Leave Job | 0 | 5
  6-Month Follow Up Interview: Very Likely to Leave Job | 1 | 5
Statistical Analysis 1: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); As the study design is quasi-experimental, there is no comparison group - both arms were analyzed jointly for each pre- and post- time interval; Test type: Other — The statistical test is a paired test assessing change at the End-of-Intervention Interview relative to baseline; p = 0.18, McNemar
Statistical Analysis 2: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 3-Month Follow Up Interview relative to baseline; p = 0.34, McNemar
Statistical Analysis 3: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 6-Month Follow Up Interview relative to baseline; p = 0.13, McNemar

2. Secondary Outcome: Change in Mean Score Over Time on Job Satisfaction Scale (JSS)
Description: Job satisfaction will be assessed using the 3-item Job Satisfaction scale (JSS). Responses are provided using a 7-point Likert scale measuring how satisfied respondents are with their job. Minimum score = 0 (worst value). Maximum score = 6 (best value). Range of scores from 0 to 18, with higher values indicating better outcomes. Measure was assessed at Baseline, at an End-of-Intervention Interview, a 3-month Follow Up Interview and at a 6-month Follow Up Interview.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Number analyzed (Participants) | 11 | 21
units on a scale
  Baseline | 15.00 (4.02) | 14.71 (3.08)
  End-of-Intervention Interview: number analyzed (Participants) | 10 | 20
  End-of-Intervention Interview | 15.80 (1.55) | 14.40 (2.14)
  3-Month Follow Up Interview: number analyzed (Participants) | 10 | 19
  3-Month Follow Up Interview | 16.20 (2.70) | 14.95 (1.87)
  6-Month Follow Up Interview: number analyzed (Participants) | 10 | 16
  6-Month Follow Up Interview | 14.00 (3.71) | 15.69 (2.44)
Statistical Analysis 1: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the End-of-Intervention Interview relative to baseline; p = 0.70, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 3-Month Follow Up Interview relative to baseline; p = 0.66, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 6-Month Follow Up Interview relative to baseline; p = 0.84, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Mean Score Over Time on Approach to Dementia Questionnaire (ADQ) - Recognition of Personhood Subscale
Description: Approach to Dementia Questionnaire (ADQ) - Recognition of Personhood Subscale is an 11-item instrument. Responses are indicated using a 5-point Likert scale. Minimum score (worst value) = 1. Maximum score (best value) = 5. Higher values represent a better outcome (range 11-55). Measure was assessed at Baseline, at an End-of-Intervention Interview, a 3-month Follow Up Interview and at a 6-month Follow Up Interview.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Number analyzed (Participants) | 11 | 21
units on a scale
  Baseline | 38.00 (3.95) | 36.86 (3.73)
  End-of-Intervention Interview: number analyzed (Participants) | 10 | 20
  End-of-Intervention Interview | 39.00 (5.25) | 38.30 (3.26)
  3-Month Follow Up Interview: number analyzed (Participants) | 10 | 19
  3-Month Follow Up Interview | 38.70 (5.66) | 37.21 (5.37)
  6-Month Follow Up Interview: number analyzed (Participants) | 10 | 16
  6-Month Follow Up Interview | 40.30 (3.83) | 38.13 (4.86)
Statistical Analysis 1: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the End-of-Intervention Interview relative to baseline; p = 0.015, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 3-Month Follow Up Interview relative to baseline; p = 0.34, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the End-of-Program Interview relative to baseline; p = 0.002, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Mean Score Over Time on Perceived Stress Scale (PSS)
Description: Perceived Stress Scale (PSS) 10-item version. Perceived stress is defined as the degree to which individuals find their lives "unpredictable, uncontrollable, and overloading". Responses are indicated using a 5-point Likert scale. Minimum score (best value)=0. Maximum score (worst value)=4. Higher values represent a worse outcome (range 0 - 40). Measure was assessed at Baseline, at an End-of-Intervention Interview, a 3-month Follow Up Interview and at a 6-month Follow Up Interview.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Number analyzed (Participants) | 11 | 21
units on a scale
  Baseline | 11.64 (4.99) | 14.19 (7.33)
  End-of-Intervention Interview: number analyzed (Participants) | 10 | 20
  End-of-Intervention Interview | 7.90 (4.38) | 12.05 (5.64)
  3-Month Follow Up Interview: number analyzed (Participants) | 10 | 19
  3-Month Follow Up Interview | 9.10 (6.67) | 11.53 (6.07)
  6-Month Follow Up Interview: number analyzed (Participants) | 10 | 16
  6-Month Follow Up Interview | 8.10 (5.61) | 12.19 (7.09)
Statistical Analysis 1: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the End-of-Intervention Interview relative to baseline; p = 0.022, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 3-Month Follow Up Interview relative to baseline; p = 0.020, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 6-Month Follow Up Interview relative to baseline; p = 0.090, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Mean Score Over Time on PROMIS Depression Scale
Description: PROMIS Emotional Distress Depression - Short Form (PROMIS) is an 8-item instrument. Responses are indicated using a 5-point Likert scale. Minimum score (best value) = 1/Never. Maximum score (worst value) = 5/Always. Lower values represent a better outcome (range 8-40). Measure was assessed at Baseline, at an End-of-Intervention Interview, a 3-month Follow Up Interview and at a 6-month Follow Up Interview.
Time Frame: Participants were followed for the duration of the intervention and 6 additional months after the intervention ends, an expected average of 8 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Number analyzed (Participants) | 11 | 21
units on a scale
  Baseline | 10.27 (2.80) | 14.29 (6.17)
  End-of-Intervention Interview: number analyzed (Participants) | 10 | 20
  End-of-Intervention Interview | 11.70 (4.27) | 11.00 (3.51)
  3-Month Follow Up Interview: number analyzed (Participants) | 10 | 19
  3-Month Follow Up Interview | 11.30 (3.47) | 11.79 (3.84)
  6-Month Follow Up Interview: number analyzed (Participants) | 10 | 16
  6-Month Follow Up Interview | 11.80 (4.21) | 12.31 (3.28)
Statistical Analysis 1: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the End-of-Intervention Interview relative to baseline; p = 0.051, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 3-Month Follow Up Interview relative to baseline; p = 0.044, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 6-Month Follow Up Interview relative to baseline; p = 1.00, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Mean Score Over Time on Maslach Burnout Inventory (MBI) - Depersonalization Subscale
Description: Burnout will be assessed via a modified Maslach Burnout Inventory (MBI) - Depersonalization Subscale (one of three subscales within the MBI), a 5-item scale. Items are measured on a 7-point Likert scale that asks how often respondents are feeling certain feelings. Minimum score (best value, never) = 0. Maximum score (worst value, every day) = 6. Analysis reports mean score rather than total score; range of the mean score is 0 to 6, with lower values representing better outcomes. Measure was assessed at Baseline, at an End-of-Intervention Interview, a 3-month Follow Up Interview and at a 6-month Follow Up Interview.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Number analyzed (Participants) | 11 | 21
units on a scale
  Baseline | 0.42 (0.56) | 0.85 (0.88)
  End-of-Intervention Interview: number analyzed (Participants) | 10 | 20
  End-of-Intervention Interview | 0.28 (0.33) | 0.59 (0.57)
  3-Month Follow Up Interview: number analyzed (Participants) | 10 | 19
  3-Month Follow Up Interview | 0.54 (0.65) | 0.72 (0.75)
  6-Month Follow Up Interview: number analyzed (Participants) | 10 | 16
  6-Month Follow Up Interview | 0.30 (0.25) | 0.61 (0.58)
Statistical Analysis 1: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the End-of-Intervention Interview relative to baseline; p = 0.023, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 3-Month Follow Up Interview relative to baseline; p = 0.56, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 6-Month Follow Up Interview relative to baseline; p = 0.16, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change in Mean Score Over Time on Maslach Burnout Inventory (MBI) - Emotional Exhaustion Subscale
Description: Burnout will be assessed via a modified Maslach Burnout Inventory (MBI) - Emotional Exhaustion Subscale (one of three subscales within the MBI), a 8-item scale. Items are measured on a 7-point Likert scale that asks how often respondents are feeling certain feelings. Minimum score (best value, never) = 0. Maximum score (worst value, every day) = 6. Analysis reports mean score rather than total score; range of the mean score is 0 to 6, with lower values representing better outcomes. Measure was assessed at Baseline, at an End-of-Intervention Interview, a 3-month Follow Up Interview and at a 6-month Follow Up Interview.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Number analyzed (Participants) | 11 | 21
units on a scale
  Baseline | 1.69 (1.13) | 2.05 (1.35)
  End-of-Intervention Interview: number analyzed (Participants) | 10 | 20
  End-of-Intervention Interview | 1.08 (0.98) | 1.84 (1.19)
  3-Month Follow Up Interview: number analyzed (Participants) | 10 | 19
  3-Month Follow Up Interview | 0.90 (0.77) | 1.91 (1.42)
  6-Month Follow Up Interview: number analyzed (Participants) | 10 | 16
  6-Month Follow Up Interview | 0.93 (0.79) | 1.58 (1.39)
Statistical Analysis 1: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the End-of-Intervention Interview relative to baseline; p = 0.15, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 3-Month Follow Up Interview relative to baseline; p = 0.12, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 6-Month Follow Up Interview relative to baseline; p = 0.018, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change in Mean Score Over Time on Maslach Burnout Inventory (MBI) - Personal Accomplishment Subscale
Description: Burnout will be assessed via a modified Maslach Burnout Inventory (MBI) - Personal Accomplishment Subscale (one of three subscales within the MBI), a 7-item scale. Items are measured on a 7-point Likert scale that asks how often respondents are feeling certain feelings. Minimum score (worst value, never) = 0. Maximum score (best value, every day) = 6. Analysis reports mean score rather than total score; range of the mean score is 0 to 6, with higher values representing better outcomes. Measure was assessed at Baseline, at an End-of-Intervention Interview, a 3-month Follow Up Interview and at a 6-month Follow Up Interview.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Number analyzed (Participants) | 11 | 21
units on a scale
  Baseline | 4.97 (0.58) | 4.59 (1.22)
  End-of-Intervention Interview | 5.07 (0.86) | 4.74 (0.95)
  3-Month Follow Up Interview: number analyzed (Participants) | 11 | 19
  3-Month Follow Up Interview | 4.99 (1.02) | 4.35 (1.12)
  6-Month Follow Up Interview: number analyzed (Participants) | 11 | 16
  6-Month Follow Up Interview | 5.14 (0.92) | 4.31 (1.25)
Statistical Analysis 1: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the End-of-Intervention Interview relative to baseline; p = 0.33, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 3-Month Follow Up Interview relative to baseline; p = 0.88, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 6-Month Follow Up Interview relative to baseline; p = 0.67, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change in Mean Score Over Time on Self-compassion Scale-Short Form (SCS-SF)
Description: The researchers will collect pre-post measures using the Self-compassion scale-short form (SCS-SF), a 12-item scale that includes the three components of self-compassion: self-kindness, common humanity, and mindfulness. This is done using a 5-point Likert scale. Minimum score = 1 (worst value). Maximum score = 5 (best value). Analysis reports mean score rather than total score (total range is 0.0 to 5.0), with higher values indicating better outcomes. Measure was assessed at Baseline, at an End-of-Intervention Interview, a 3-month Follow Up Interview and at a 6-month Follow Up Interview.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Number analyzed (Participants) | 11 | 21
units on a scale
  Baseline | 3.72 (0.52) | 2.73 (0.38)
  End-of-Intervention Interview: number analyzed (Participants) | 10 | 20
  End-of-Intervention Interview | 3.64 (0.61) | 3.77 (0.58)
  3-Month Follow Up Interview: number analyzed (Participants) | 10 | 19
  3-Month Follow Up Interview | 3.71 (0.50) | 3.88 (0.62)
  6-Month Follow Up Interview: number analyzed (Participants) | 10 | 16
  6-Month Follow Up Interview | 3.68 (0.34) | 3.85 (0.66)
Statistical Analysis 1: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the End-of-Intervention Interview relative to baseline; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 3-Month Follow Up Interview relative to baseline; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 6-Month Follow Up Interview relative to baseline; p < 0.001, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change in Mean Score Over Time on Self-compassion Scale-Short Form (SCS-SF) - Self-kindness Subscale
Description: The researchers will collect pre-post measures using the Self-compassion scale-short form (SCS-SF) - Self-kindness Subscale (one of six subscales within the SCS-SF), a 3-item scale. Items are measured on a 5-point Likert scale. Minimum score = 1 (worst value). Maximum score = 5 (best value), higher scores indicating better outcomes. Analysis reports mean score rather than total score (total range is 0.0 to 5.0). Measure was assessed at Baseline, at an End-of-Intervention Interview, a 3-month Follow Up Interview and at a 6-month Follow Up Interview.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Number analyzed (Participants) | 11 | 21
units on a scale
  Baseline | 4.00 (0.75) | 3.22 (0.61)
  End-of-Intervention Interview: number analyzed (Participants) | 10 | 20
  End-of-Intervention Interview | 3.50 (0.96) | 3.75 (0.73)
  3-Month Follow Up Interview: number analyzed (Participants) | 10 | 19
  3-Month Follow Up Interview | 3.80 (1.12) | 3.84 (0.61)
  6-Month Follow Up Interview: number analyzed (Participants) | 10 | 16
  6-Month Follow Up Interview | 3.87 (0.69) | 3.90 (0.80)
Statistical Analysis 1: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the End-of-Intervention Interview relative to baseline; p = 0.17, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 3-Month Follow Up Interview relative to baseline; p = 0.020, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 6-Month Follow Up Interview relative to baseline; p = 0.062, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change in Mean Score Over Time on Self-compassion Scale-Short Form (SCS-SF) - Self-judgment Subscale
Description: The researchers will collect pre-post measures using the Self-compassion scale-short form (SCS-SF) - Self-judgment Subscale (one of six subscales within the SCS-SF), a 3-item scale. Items are measured on a 5-point Likert scale. Minimum score = 1 (best value). Maximum score = 5 (worst value), with lower scores indicating better outcomes. Analysis reports mean score rather than total score (total range is 0.0 to 5.0). Measure was assessed at Baseline, at an End-of-Intervention Interview, a 3-month Follow Up Interview and at a 6-month Follow Up Interview.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Number analyzed (Participants) | 11 | 21
units on a scale
  Baseline | 2.39 (0.96) | 3.33 (0.99)
  End-of-Intervention Interview: number analyzed (Participants) | 10 | 20
  End-of-Intervention Interview | 2.43 (1.31) | 2.25 (0.89)
  3-Month Follow Up Interview: number analyzed (Participants) | 10 | 19
  3-Month Follow Up Interview | 2.20 (0.80) | 1.95 (0.86)
  6-Month Follow Up Interview: number analyzed (Participants) | 10 | 16
  6-Month Follow Up Interview | 2.13 (0.50) | 2.08 (0.82)
Statistical Analysis 1: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the End-of-Intervention Interview relative to baseline; p = 0.013, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 3-Month Follow Up Interview relative to baseline; p = 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 6-Month Follow Up Interview relative to baseline; p = 0.003, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Change in Mean Score Over Time on Self-compassion Scale-Short Form (SCS-SF) - Common Humanity Subscale
Description: The researchers will collect pre-post measures using the Self-compassion scale-short form (SCS-SF) - Common humanity Subscale (one of six subscales within the SCS-SF), a 3-item scale. Items are measured on a 5-point Likert scale. Minimum score = 1 (worst value). Maximum score = 5 (best value), with higher scores indicating better outcomes. Analysis reports mean score rather than total score (total range is 0.0 to 5.0). Measure was assessed at Baseline, at an End-of-Intervention Interview, a 3-month Follow Up Interview and at a 6-month Follow Up Interview.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Number analyzed (Participants) | 11 | 21
units on a scale
  Baseline | 3.48 (0.85) | 2.56 (0.99)
  End-of-Intervention: number analyzed (Participants) | 10 | 20
  End-of-Intervention | 3.83 (0.76) | 3.67 (0.84)
  3-Month Follow Up Interview: number analyzed (Participants) | 10 | 19
  3-Month Follow Up Interview | 3.37 (1.21) | 3.68 (0.86)
  6-Month Follow Up Interview: number analyzed (Participants) | 10 | 16
  6-Month Follow Up Interview | 3.03 (0.67) | 3.63 (1.13)
Statistical Analysis 1: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the End-of-Intervention Interview relative to baseline; p = 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 3-Month Follow Up Interview relative to baseline; p = 0.010, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 6-Month Follow Up Interview relative to baseline; p = 0.085, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Change in Mean Score Over Time on Self-compassion Scale-Short Form (SCS-SF) - Isolation Subscale
Description: The researchers will collect pre-post measures using the Self-compassion scale-short form (SCS-SF) - Isolation Subscale (one of six subscales within the SCS-SF), a 3-item scale. Items are measured on a 5-point Likert scale. Minimum score = 1 (best value). Maximum score = 5 (worst value), with lower scores indicating better outcomes. Analysis reports mean score rather than total score (total range is 0.0 to 5.0). Measure was assessed at Baseline, at an End-of-Intervention Interview, a 3-month Follow Up Interview and at a 6-month Follow Up Interview.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Number analyzed (Participants) | 11 | 21
units on a scale
  Baseline | 2.55 (0.95) | 3.41 (0.55)
  End-of-Intervention: number analyzed (Participants) | 10 | 20
  End-of-Intervention | 2.37 (0.94) | 2.18 (0.88)
  3-Month Follow Up Interview: number analyzed (Participants) | 10 | 19
  3-Month Follow Up Interview | 2.20 (0.77) | 1.91 (0.83)
  6-Month Follow Up Interview: number analyzed (Participants) | 10 | 16
  6-Month Follow Up Interview | 2.23 (0.88) | 1.85 (0.75)
Statistical Analysis 1: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the End-of-Intervention Interview relative to baseline; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 3-Month Follow Up Interview relative to baseline; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 6-Month Follow Up Interview relative to baseline; p < 0.001, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Change in Mean Score Over Time on Self-compassion Scale-Short Form (SCS-SF) - Mindfulness Subscale
Description: The researchers will collect pre-post measures using the Self-compassion scale-short form (SCS-SF) - Mindfulness Subscale (one of six subscales within the SCS-SF), a 3-item scale. Items are measured on a 5-point Likert scale. Minimum score = 1 (worst value). Maximum score = 5 (best value), with higher scores indicating better outcomes. Analysis reports mean score rather than total score (total range is 0.0 to 5.0). Measure was assessed at Baseline, at an End-of-Intervention Interview, a 3-month Follow Up Interview and at a 6-month Follow Up Interview.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Number analyzed (Participants) | 11 | 21
units on a scale
  Baseline | 4.24 (0.72) | 2.68 (1.06)
  End-of-Intervention Interview: number analyzed (Participants) | 10 | 20
  End-of-Intervention Interview | 3.83 (0.77) | 3.77 (0.77)
  3-Month Follow Up Interview: number analyzed (Participants) | 10 | 19
  3-Month Follow Up Interview | 3.53 (0.82) | 3.84 (0.83)
  6-Month Follow Up Interview: number analyzed (Participants) | 10 | 16
  6-Month Follow Up Interview | 3.80 (0.96) | 3.77 (0.79)
Statistical Analysis 1: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the End-of-Intervention Interview relative to baseline; p = 0.046, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 3-Month Follow Up Interview relative to baseline; p = 0.14, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 6-Month Follow Up Interview relative to baseline; p = 0.058, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Change in Mean Score Over Time on Self-compassion Scale-Short Form (SCS-SF) - Over-identification Subscale
Description: The researchers will collect pre-post measures using the Self-compassion scale-short form (SCS-SF) - Over-identification Subscale (one of six subscales within the SCS-SF), a 3-item scale. Items are measured on a 5-point Likert scale. Minimum score = 1 (best value). Maximum score = 5 (worst value), with lower scores indicating better outcomes. Analysis reports mean score rather than total score (total range is 0.0 to 5.0). Measure was assessed at Baseline, at an End-of-Intervention Interview, a 3-month Follow Up Interview and at a 6-month Follow Up Interview.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Number analyzed (Participants) | 11 | 21
units on a scale
  Baseline | 2.45 (1.00) | 3.32 (0.45)
  End-of-Intervention Interview: number analyzed (Participants) | 10 | 20
  End-of-Intervention Interview | 2.53 (0.98) | 2.15 (0.83)
  3-Month Follow Up Interview: number analyzed (Participants) | 10 | 19
  3-Month Follow Up Interview | 2.07 (0.60) | 2.25 (0.86)
  6-Month Follow Up Interview: number analyzed (Participants) | 10 | 16
  6-Month Follow Up Interview | 2.27 (0.44) | 2.23 (0.97)
Statistical Analysis 1: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the End-of-Intervention Interview relative to baseline; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 3-Month Follow Up Interview relative to baseline; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: 8-Week Mindful Self-Compassion (MSC) vs 6-Week Mindful Self Compassion (MSC); [analysis description as in outcome 1, analysis 1]; Test type: Other — The statistical test is a paired test assessing change at the 6-Month Follow Up Interview relative to baseline; p < 0.001, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Percent of Classes Attended by Participating CNAs
Description: This will be reported as percent of classes attended by CNAs.
Time Frame: Participants will be followed for the duration of the intervention, an expected average of 6-8 weeks
Population: Analysis population is composed of participants who completed the 6/8-week intervention. All collected data are reported. Some data are missing due to study attrition or nonresponse.
Measure: Number; unit: percentage of classes attended by CNAs
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Number analyzed (Participants) | 10 | 20
percentage of classes attended by CNAs | 93.75 | 95.67

17. Secondary Outcome: Percent of Participants Attending All Intervention Sessions
Description: This will be reported by percent of participants who attended every assigned intervention session (6 or 8 depending on intervention arm).
Time Frame: Participants will be followed for the duration of the intervention, an expected average of 6-8 weeks
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Number analyzed (Participants) | 10 | 20
percentage of participants | 50.00 | 75.00

18. Secondary Outcome: Percent Intervention Minutes Attended by Participants
Description: This will be collected by recording the number of minutes each participant spent per class in order to account for intervention missed due to participants' leaving early or coming late, and reporting percent of minutes attended by participants.
Time Frame: Participants will be followed for the duration of the intervention, an expected average of 6-8 weeks
Population: as for outcome 16
Measure: Number; unit: percentage of intervention minutes
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Number analyzed (Participants) | 10 | 20
percentage of intervention minutes | 95.35 | 98.17

19. Secondary Outcome: Mean Number of Days Per Week Spent in Out-of-Class Informal Exercise
Description: Based on participant completion of weekly surveys, the researchers will measure the number of days each week that class participants were able to practice learned informal techniques and exercises outside of class hours.
Time Frame: Participants will be followed for the duration of the intervention, an expected average of 6/8 weeks
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: days a week
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Number analyzed (Participants) | 10 | 20
days a week | 2.58 (1.25) | 2.60 (1.10)

20. Secondary Outcome: Mean Number of Days Per Week Spent in Out-of-Class Formal Exercise
Description: Based on participant completion of weekly surveys, the researchers will measure the number of days each week that class participants were able to practice learned formal techniques and exercises outside of class hours.
Time Frame: Participants will be followed for the duration of the intervention, an expected average of 6/8 weeks
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: days a week
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Number analyzed (Participants) | 10 | 20
days a week | 2.12 (1.56) | 2.60 (2.47)

21. Secondary Outcome: Study Participant's Self-Rating of Satisfaction With the MSC Course
Description: The researchers assess satisfaction of the MSC training using an 8-item, 5-point Likert Scale (0 = Strongly Disagree, 1 = Disagree, 2 = Neither Agree nor Disagree, 3 = Agree, 4 = Strongly Agree). Minimum = 0 (worst value), maximum = 4 (best value). Measure was assessed during the End-of-Intervention Interview.
Time Frame: At the conclusion of the week 6/8 class, during the End-of-Intervention Interview, participants were asked their satisfaction with the course
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
Number analyzed (Participants) | 10 | 20
Participants
  I was satisfied with the course.: Strongly Disagree | 0 | 0
  I was satisfied with the course.: Disagree | 0 | 0
  I was satisfied with the course.: Neither Agree nor Disagree | 0 | 0
  I was satisfied with the course.: Agree | 0 | 1
  I was satisfied with the course.: Strongly Agree | 10 | 19
  The length for each class session was just the right amount of time.: Strongly Disagree | 0 | 1
  The length for each class session was just the right amount of time.: Disagree | 1 | 1
  The length for each class session was just the right amount of time.: Neither Agree nor Disagree | 1 | 2
  The length for each class session was just the right amount of time.: Agree | 4 | 12
  The length for each class session was just the right amount of time.: Strongly Agree | 4 | 4
  Having a class session once a week was just the right amount of sessions per week.: Strongly Disagree | 0 | 0
  Having a class session once a week was just the right amount of sessions per week.: Disagree | 1 | 0
  Having a class session once a week was just the right amount of sessions per week.: Neither Agree nor Disagree | 0 | 2
  Having a class session once a week was just the right amount of sessions per week.: Agree | 5 | 5
  Having a class session once a week was just the right amount of sessions per week.: Strongly Agree | 4 | 13
  I intend to use the skills I learned in this course.: Strongly Disagree | 0 | 0
  I intend to use the skills I learned in this course.: Disagree | 0 | 0
  I intend to use the skills I learned in this course.: Neither Agree nor Disagree | 0 | 0
  I intend to use the skills I learned in this course.: Agree | 2 | 1
  I intend to use the skills I learned in this course.: Strongly Agree | 8 | 19
  Taking this course has made a difference in my work life.: Strongly Disagree | 0 | 0
  Taking this course has made a difference in my work life.: Disagree | 0 | 0
  Taking this course has made a difference in my work life.: Neither Agree nor Disagree | 0 | 0
  Taking this course has made a difference in my work life.: Agree | 1 | 7
  Taking this course has made a difference in my work life.: Strongly Agree | 9 | 13
  Taking this course has made a difference in my personal life.: Strongly Disagree | 0 | 0
  Taking this course has made a difference in my personal life.: Disagree | 0 | 0
  Taking this course has made a difference in my personal life.: Neither Agree nor Disagree | 0 | 0
  Taking this course has made a difference in my personal life.: Agree | 2 | 8
  Taking this course has made a difference in my personal life.: Strongly Agree | 8 | 12
  I would suggest this course to a friend.: Strongly Disagree | 0 | 0
  I would suggest this course to a friend.: Disagree | 0 | 0
  I would suggest this course to a friend.: Neither Agree nor Disagree | 0 | 0
  I would suggest this course to a friend.: Agree | 2 | 1
  I would suggest this course to a friend.: Strongly Agree | 8 | 19
  I find this course to be useful in my daily life.: Strongly Disagree | 0 | 0
  I find this course to be useful in my daily life.: Disagree | 0 | 0
  I find this course to be useful in my daily life.: Neither Agree nor Disagree | 0 | 0
  I find this course to be useful in my daily life.: Agree | 1 | 3
  I find this course to be useful in my daily life.: Strongly Agree | 9 | 17

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the course of the intervention and follow-up interviews. This total time period was 8 months per participant.
Groups:
- 8-Week Mindful Self-Compassion (MSC): CNAs in Aim 1 will participate in the standardized, 8-week Mindful Self-Compassion course. Each 8-week session will last for 2.5 hours. Also included is a half day retreat, that CNAs may attend if they are able.
  8-Week Mindful Self-Compassion (MSC): The 8-week MSC is a course of eight 2.5 hour weekly sessions that is based off self-compassion, a construct closely related to mindfulness. Self-compassion (SC) has three main interrelated components: self-kindness, common humanity, and mindfulness. MSC is an 8-session program that integrates SC and mindfulness.
  It includes the following components:
  * Discovering Mindful Self-Compassion
  * Practicing Mindfulness
  * Practicing Lovingkindness
  * Discovering your Compassionate Voice
  * Living Deeply
  * Meeting Difficult Emotions
  * Exploring Challenging Relationships
  * Embracing Your Life
Arm/Group | 8-Week Mindful Self-Compassion (MSC) | 6-Week Mindful Self Compassion (MSC)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/11 | 1/21
Other Adverse Events (participants affected / at risk) | 0/11 | 1/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8-Week Mindful Self-Compassion (MSC) (N=11) | 6-Week Mindful Self Compassion (MSC) (N=21)
Vehicular Accident (Surgical and medical procedures) | 0 (0) | 1 (1) — Participant reported a vehicular accident after the end-of-intervention, during 3-month Follow Up Interview.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8-Week Mindful Self-Compassion (MSC) (N=11) | 6-Week Mindful Self Compassion (MSC) (N=21)
Pulled Muscle (Infections and infestations) | 0 (0) | 1 (1) — Participant pulled a side muscle at during work.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT03720652/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/52/NCT03720652/SAP_001.pdf